CLINICAL TRIAL: NCT04739995
Title: 12-month Randomized, Double-blind, Placebo-controlled, Pharmacological Clinical Trial to Evaluate the Effectiveness, Cost-utility and Neurobiological Effects of Low-dose Naltrexone in Patients With Fibromyalgia (INNOVA Project)
Brief Title: Cost-utility and Physiological Effects of LDN in Patients With Fibromyalgia
Acronym: INNOVA
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICI20/00080
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Randomized Controlled Trial
MeSH Terms: interventions — Naltrexone

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Dose-Naltrexone (LDN) (Experimental): The LDN treatment will consist of one 4.5 mg naltrexone tablet (lactose-free) taken daily for 12 months before going to sleep.
  Interventions: Drug: Low-dose naltrexone
- Placebo (Placebo Comparator): The control group will take the placebo daily (a film-coated tablet, identical to the LDN, filled with a lactose-free excipient), for 12 months, following the same guidelines.
  Interventions: Drug: Low-dose naltrexone

INTERVENTIONS:
Drug: Low-dose naltrexone — 4.5 mg LDN/day for 1 year
  Other Names: LDN

SUMMARY:
Background: Low-dose naltrexone (LDN) may be useful in managing the pathologies that alter inflammatory markers, such as Crohn's disease or fibromyalgia (FM). The anti-inflammatory effect of LDN should be produced through the inhibition of Toll-like receptor 4 activity expressed in the membrane of various immune system cells (e.g. microglia). Conversely, due to a rebound effect, LDN could exercise an analgesic effect that strengthens the endogenous inhibitory system. According to this hypothesis, the low-intensity and intermittent blocking of the opioid receptors generated by LDN should induce a compensatory mechanism that should facilitate an increase in the production of endogenous opioids and greater sensitivity of the system to their effects. To date, the effects of LDN in patients with FM have been evaluated through crossover studies that have yielded promising results. Given that the studies conducted up to now have had small sample sizes and crossover designs, and given that there are still no studies in which its potential cost-utility is assessed, studies with greater methodological rigor and larger samples are necessary to confirm the effectiveness of LDN in FM.

Jointly evaluating the effectiveness and cost-utility, the changes in metabolites in certain areas of the brain, and systemic inflammatory markers potentially linked to the etiopathogenesis of FM, should allow us to gain a more detailed knowledge of the neurobiological mechanisms underlying the effectiveness of LDN in this population.

Objectives: To evaluate the effectiveness and safety of LDN in patients with FM and analyse its cost-utility both from the government and the healthcare perspective at 1-year follow-up. Brain metabolites and systemic inflammatory biomarkers will be included to evaluate neurobiological mechanisms behind LDN therapeutic effects.

Design: Randomized, Controlled Trial. Centre: Parc Sanitari Sant Joan de Déu (St. Boi de Llobregat, Spain). Participants: 120 patients with FM will be randomly assigned to LDN (4.5mg/day) or placebo.

Main outcome measure: Pain severity using Ecological Momentary Assessment. Secondary outcomes: functionality, affective symptoms, fibrofog, quality of life. Costs and QALYs will be also calculated. Biomarkers: 50% of the patients will be scanned at baseline and at week 12 for changes in brain metabolites related to neuroinflammation and central sensitization. Immune-inflammatory markers in serum will also be evaluated.

DETAILED DESCRIPTION:
Low-dose Naltrexone (LDN): A potential treatment for fibromyalgia (FM)

Naltrexone is an opioid antagonist used for treating opiate and alcohol dependency that blocks the mu receptors and, to a lesser extent, the delta-opioid receptors. There is growing evidence that naltrexone administered in very low doses (i.e. low-dose naltrexone, LDN) -approximately 1/10 of the usual dose, between 1.5-5 mg vs. 50 mg/day- may be useful in managing the various pathologies that alter inflammatory markers, such as Crohn's disease, multiple sclerosis and FM.

The anti-inflammatory effect of naltrexone should be produced through the inhibition of TLR-4 (Toll-like receptor 4) activity expressed in the membrane of various immune system cells (e.g. microglia, macrophages). Conversely, due to a "rebound effect", LDN could exercise an analgesic effect that strengthens the endogenous inhibitory system. According to this hypothesis, the low-intensity and intermittent blocking of the opioid receptors generated by LDN should induce a compensatory mechanism that should facilitate an increase in the production of endogenous opioids and greater sensitivity of the system to their effects. To date, the effects of LDN in patients with FM have only been evaluated through crossover pilot studies and have always produced highly promising results. Thus, in the first study conducted with LDN in FM (N= 10), ameliorations in the daily pain, stress and fatigue levels were observed. In the same vein, in a posterior study (N= 31), significant improvements (vs. Placebo) in daily pain (28% vs. 18%), satisfaction with life and mood were also observed. In another single-blind crossover study (N= 8) the pre and post changes in the levels of cytokines in plasma were evaluated over 8 weeks, with reductions in a wide range of inflammatory markers being observed (e.g. IL-1, sIL-1ra, IL-6, IL-10, TNF-alpha), as well as changes in the levels of pain (-15%) and FM symptoms (-18%). Given that the studies conducted up to now had reduced sample sizes and crossover designs, and given that there are still no studies in which its potential cost-utility is assessed, studies with greater methodological rigor and larger samples are necessary to confirm the clinical effectiveness of LDN in FM. Jointly evaluating the efficacy and cost-utility analyses, the changes in metabolites (i.e. Glu) in certain areas of the brain, and systemic inflammatory markers potentially linked to the etiopathogenesis of FM, should allow us to gain a more detailed knowledge of the neurobiological mechanisms underlying the effectiveness of LDN in this population. The INNOVA project will enable all these factors to be evaluated for the first time.

ELIGIBILITY:
General Inclusion Criteria:

* Female between 18 and 70 years old
* Patients diagnosed of FM according to ACR 2016 criteria
* Chronic widespread pain for at least 6 months ranked ≥ 4 out of 10;
* Understand Spanish;
* Written informed written consent;

General Exclusion Criteria:

* Treatment with opiates in last 3 months;
* Diagnosis of severe medical/psychiatric disorders (e.g. cancer, severe depression, psychotic disorder, schizophrenia);
* Being pregnant (or planning a pregnancy during the study period) or breastfeeding;
* Known allergy to naltrexone or naloxone;
* Hematological disorders;
* Abnormal hepatic function;
* Taking anticoagulant medication;
* Alcohol consume during the study period
* Participation in other clinical trials;

Additional inclusion criteria for biomarker sub-study:

Right-handed (for the neuroimaging tests)

Additional exclusion criteria for biomarker sub-study:

Comorbid rheumatologic illnesses (e.g. rheumatoid arthritis, lupus); fever (> 38ºC) or infection in the last 2 weeks; vaccination in the last 4 weeks; Take drugs with anti-inflammatory effects in the 72h prior to blood / neuroimaging; taking cortisone or anti-cytokine therapy; needle phobia; inability to be scanned (due to claustrophobia, metal implants, pacemakers, etc.); Body Mass Index (BMI) > 36 kg/m2; consumption of > 8 units of caffeine per day; smoking > 10 cigarettes/day; acute pain not-related to FM on the day of the scan (e.g. headache, back pain).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 99 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Through study completion, an average of 1 year
  -Numerical Rating Scale-NRS- from 0 (no pain) to 10 (worst possible pain)

SECONDARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire (FIQR) | Through study completion, an average of 1 year
  21-item questionnaire on physical function, overall impact and severity of the symptoms associated with FM. Total scores can range from 0 (no impairment) to (maximum impairment) memory/attentional problems, quality of sleep)
Depression Anxiety Stress Scale (DASS-21) | Through study completion, an average of 1 year
  Scale of 21 items created to assess symptoms of depression, anxiety and stress. Each subscale (Depressión, Anxiety and Stress) includes 7 items with scores ranging from 0 to 21. Higher scores indicate higher symptom severity.
Multidimensional Inventory of Subjective Cognitive Impairment (MISCI) | Through study completion, an average of 1 year
  10-item measure of subjective cognitive dysfunction in FM. total score ranges from 10 to 50, where lower scores indicate higher cognitive dysfunction.

OTHER OUTCOMES:
EuroQoL (EQ-5D-5L) | Through study completion, an average of 1 year
  Instrument for evaluating health-related quality of life. The EQ-5D-5L scores will be used to calculate the QualityAdjusted Life Years (QALYs) for the cost-utility analysis
Client Service Receipt Inventory (CSRI) | Through study completion, an average of 1 year
  The version used in this study is designed to retrospectively collect information on the use of health and social services during the previous 12 months. This instrument does not provide total or sub-scale scores, only collects information about use of services and medication consumption.
Patient Global and Specific Impression of Change (PGIC/PSIC) | Through study completion, an average of 1 year
  Items scored on a 7-point Likert scale (from 1 "much better" to 7 "much worse")
ACTTION AE | Through study completion, an average of 1 year
  It is a reporting checklist used to measure safety and benefit-risk of a clinical trial.
The Pain Monitor® app | Through study completion, an average of 1 year
  It was validated in an empirical study for use on Android smartphones. It will be used to assess daily (twice a day) the level of pain, fatigue, etc. during the treatment period.
Socio-demographic questionnaire | Baseline
  Gender, date of birth, marital status, living arrangements, educational level and work status.
12-item WHODAS 2.0 | Baseline
  The 12-item interviewer administered version of the World Health Organization Disability Assessment Schedule 2.0 can be used algorithmically for the probable diagnosis of a depressive disorder, or as a continuous measure of scores ranging from 0 to 27, with cutoff points of 5, 10, 15 and 20, which set the levels of symptoms of depression as mild, moderate, moderately severe or severe.
Generalized Anxiety Disorder 7-item scale (GAD-7) | Baseline
  Questionnaire that measures generalized anxiety symptoms (pathological worry). This instrument has been used in other studies for FM.
Fibromyalgia Survey Diagnostic Criteria (FSDC) | Baseline
  Scale that assesses the main symptoms of FM according to the latest revision of the American College of Rheumatology (ACR) criteria. This instrument includes 2 subscales: (1) the generalized pain index and (2) the symptom severity scale. A total FM score is obtained, with higher values indicating greater severity (range: 0 to 31 points).

CONTACTS AND LOCATIONS:
Overall Officials: Juan V. Luciano, PhD, Principal Investigator — Fundació Sant Joan de Déu
Locations (1):
- Parc Sanitari Sant Joan de Déu (PSSJD), Sant Boi de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colomer-Carbonell A, Sanabria-Mazo JP, Hernandez-Negrin H, Borras X, Suso-Ribera C, Garcia-Palacios A, Muchart J, Munuera J, D'Amico F, Maes M, Younger JW, Feliu-Soler A, Rozadilla-Sacanell A, Luciano JV. Study protocol for a randomised, double-blinded, placebo-controlled phase III trial examining the add-on efficacy, cost-utility and neurobiological effects of low-dose naltrexone (LDN) in patients with fibromyalgia (INNOVA study). BMJ Open. 2022 Jan 6;12(1):e055351. doi: 10.1136/bmjopen-2021-055351. PMID 34992118